CLINICAL TRIAL: NCT07310693
Title: External Validation of a Predictive Model for Occult Cancer Risk in Patients With Venous Thromboembolism Developed Using Machine Learning
Brief Title: External Validation of the CLOVER Score for Detecting Occult Cancer in Venous Thromboembolism Patients
Acronym: CLOVER
Status: Recruiting | Type: Observational
Sponsor: Infanta Leonor University Hospital (Other)
Collaborators: Fundación para la Investigación e Innovación Biomédica del Hospital Universitario Infanta Leonor (Unknown)
Responsible Party: Principal Investigator, Anabel Franco Moreno, Specialist in Internal Medicine, Infanta Leonor University Hospital
Other Study IDs: CLOVER_validation
Record Dates: First submitted 2025-12-08; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism (VTE); Occult Cancer
Keywords: Occult Cancer; Venous thromboembolism; Machine learning; Prediction model; External validation; CLOVER score
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective VTE Cohort: Adults with objectively confirmed symptomatic venous thromboembolism (deep vein thrombosis and/or pulmonary embolism) consecutively enrolled from December 2025 to December 2027 in participating hospitals. All participants will undergo routine clinical evaluation, laboratory testing, and cancer screening according to standard practice. The CLOVER score will be calculated at baseline using the web-based tool (CLOVER-Web).

SUMMARY:
This study aims to externally validate the CLOVER score, a machine learning-based predictive model designed to identify patients with venous thromboembolism (VTE) who are at increased risk of having an occult cancer. The study includes a retrospective cohort of patients with acute symptomatic VTE diagnosed between 2000 and 2022, and a prospective cohort of consecutively recruited patients from December 2025 to December 2027. The CLOVER model will be applied to all participants, and its ability to discriminate between patients with and without occult cancer will be evaluated. The study also assesses clinicians' satisfaction with the web-based tool (CLOVER-Web) developed to facilitate the use of the score in clinical practice.

DETAILED DESCRIPTION:
This study aims to externally validate the CLOVER score, a machine learning-based predictive model designed to identify patients with venous thromboembolism (VTE) who are at increased risk of having an occult cancer. The study combines a retrospective and a prospective cohort.

Retrospective cohort:

Patients aged ≥18 years with objectively confirmed symptomatic deep vein thrombosis (DVT) and/or pulmonary embolism (PE) diagnosed between January 1, 2000, and August 31, 2022, in participating hospitals across Spain will be included. Patients from centers involved in the model derivation (Hospital Universitario Infanta Leonor and Hospital Universitario de Fuenlabrada) will be excluded. Cases are defined as patients with a histologically confirmed cancer diagnosis occurring between 1 and 24 months after the index VTE event. Controls are defined as patients without a cancer diagnosis during the same period. All variables required for the CLOVER model (age, D-dimer, systolic blood pressure, ALT, hemoglobin, creatinine, total cholesterol, platelet count, triglycerides, leukocyte count, weight, chronic lung disease, heart rate, sex, and previous VTE recurrence) will be extracted from electronic health records using a standardized data collection form. The CLOVER model will be applied to each patient to assess its discrimination for cancer prediction in the retrospective cohort.

Prospective cohort:

From December 1, 2025, to December 31, 2027, consecutive adult patients with objectively confirmed symptomatic VTE will be recruited in participating hospitals. All patients will undergo a standard clinical evaluation including medical history, physical examination, basic laboratory testing (complete blood count and biochemistry), chest X-ray, and age- and sex-appropriate cancer screening tests according to clinical practice guidelines. The CLOVER score will be calculated at the time of VTE diagnosis using a dedicated web-based tool (CLOVER-Web). Patients will be classified as "low risk" or "high risk" based on the optimal F1-score threshold (0.487), corresponding to a sensitivity of 51%, specificity of 95%, PPV of 46%, and NPV of 96%. All participants will be followed for at least two years to determine whether an occult cancer is diagnosed. Further diagnostic testing for suspected cancer will be performed at the discretion of the treating physician, regardless of CLOVER result.

Model performance and bias assessment:

The external validation will evaluate model discrimination using sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and the area under the ROC curve (AUC). Additional analyses will assess potential prediction bias across demographic and clinical subgroups (e.g., age, sex, comorbidities). Model calibration and temporal performance will also be reviewed, with predefined procedures for identifying deviations from expected behavior. Weekly reports during the prospective phase will alert investigators to performance drift or potential implementation issues in the web-based tool.

Clinician satisfaction:

A secondary objective is to evaluate clinician satisfaction with the CLOVER-Web tool. An online questionnaire specifically designed for this study will be administered to participating clinicians to assess usability, clarity, and clinical utility.

Ethical considerations:

The study follows the Declaration of Helsinki and Spanish regulations on biomedical research and data protection. Retrospective data collection will request exemption from informed consent due to the use of anonymized clinical information. Prospective participants will provide written or electronic informed consent. All data will be pseudonymized and stored securely.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Objectively confirmed acute symptomatic venous thromboembolism (deep vein thrombosis and/or pulmonary embolism).
* Ability to provide written or electronic informed consent.

Exclusion Criteria:

* Suspicion of cancer during the initial diagnostic evaluation for VTE.
* Participation in another interventional study that may interfere with outcomes.
* Inability or refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with objectively confirmed symptomatic venous thromboembolism (deep vein thrombosis or pulmonary embolism) who are consecutively recruited in participating hospitals in Spain. All participants undergo routine clinical evaluation, laboratory testing, and age- and sex-appropriate cancer screening according to standard practice. The population represents real-world patients with new-onset VTE without known or suspected cancer at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of occult cancer within 24 months | 24 months
  Proportion of participants with a histologically confirmed diagnosis of occult cancer identified between 1 and 24 months after the index venous thromboembolism (VTE) event. Occult cancer is defined as a new cancer diagnosis not clinically evident at the time of VTE diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Anabel Franco-Moreno, MD, PhD, Principal Investigator — Hospital Universitario Infanta Leonor; Franco-Moreno, MD, PhD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (12):
- Spain (12):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid, Madrid
  - Hospital Universitatio del Sureste, Madrid, Madrid
  - Hospital Universitario de Móstoles, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario Morales Meseguer, Murcia, Murcia
  - Hospital San Agustín, Avilés, Principality of Asturias
  - Hospital Universitario Son Llatzer, Balea
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including baseline characteristics, clinical variables, imaging results, and outcomes related to occult cancer detection. Data will be made available to qualified investigators upon reasonable request and after signing a data sharing agreement ensuring confidentiality and appropriate use. IPD will be available beginning 12 months after study completion and will remain accessible for 5 years. Access to IPD will be granted to qualified researchers with a methodologically sound research proposal. Requests must be submitted to the study's coordinating center and will be evaluated by the principal investigators. A data use agreement will be required before any data transfer. Data will be hosted on the HORUS-ML secure research platform (restricted access).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning 12 months after the completion of the study and will remain accessible for a period of 5 years. Supporting documentation will be provided during the same availability window.
Access Criteria: IPD will be available to qualified researchers who submit a methodologically sound research proposal. All requests must be evaluated and approved by the principal investigators. Access will require signing a data use agreement ensuring confidentiality and appropriate use. Data will be shared through the secure HORUS-ML platform.

REFERENCES:
- [Background] Franco-Moreno A, Madronal-Cerezo E, de Ancos-Aracil CL, Farfan-Sedano AI, Munoz-Rivas N, Bascunana Morejon-Giron J, Ruiz-Giardin JM, Alvarez-Rodriguez F, Prada-Alonso J, Gala-Garcia Y, Casado-Suela MA, Bustamante-Fermosel A, Alfaro-Fernandez N, Torres-Macho J; CLOVER Research Group. Development of a Predictive Model of Occult Cancer After a Venous Thromboembolism Event Using Machine Learning: The CLOVER Study. Medicina (Kaunas). 2024 Dec 27;61(1):18. doi: 10.3390/medicina61010018. PMID 39859000